CLINICAL TRIAL: NCT06812208
Title: Implementation Strategies to Decentralize Breast Ultrasound Services and Facilitate Timely Breast Cancer Diagnoses in Rwanda
Brief Title: Strategies to Decentralize Breast Ultrasound in Rwanda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners in Health (Other); Memorial Sloan Kettering Cancer Center (Other); University of Pennsylvania (Other); Harvard Medical School (HMS and HSDM) (Other); Obafemi Awolowo University (Other); Kaiser Permanente (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lydia Pace, MD, MPH, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024P002311
Record Dates: First submitted 2025-01-25; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Early Detection of Cancer; Ultrasonography
Keywords: breast ultrasound; implementation strategies; low and middle income countries; breast cancer early detection; teleultrasound; Rwanda
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Type 2 hybrid implementation-effectiveness study designed to compare the effect of synchronous teleultrasound mentorship versus asynchronous virtual feedback (implementation strategies) on penetration of breast ultrasound into district hospital practice (implementation outcome) and ultrasound quality (clinical outcome).
Who Masked: Outcomes Assessor
Masking Description: The research team members who are evaluating the strategies will not know which district hospitals belong to each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teleultrasound (Experimental): Arm 1 hospitals will receive teleultrasound supervision using secure Reacts software which allows clinical supervisors to view ultrasound images and provide scanning feedback in real-time.
  Interventions: Behavioral: Teleultrasound with Philips Lumify ultrasound probes and Reacts software
- Asynchronous virtual feedback (Active Comparator): Arm 2 hospitals will receive asynchronous virtual feedback in which trainees will upload static images to a shared drive and mentors will email feedback within 24 hours.
  Interventions: Behavioral: Asynchronous virtual feedback

INTERVENTIONS:
Behavioral: Teleultrasound with Philips Lumify ultrasound probes and Reacts software — Clinicians at hospitals randomized to Arm 1 will be provided with Reacts licenses and trained to use Reacts with Philips Lumify devices immediately following the baseline training. Each hospital will be assigned to 2-3 radiologist supervisors (typically 1 Rwandan, 1 U.S.-based), with at least one available on each designated U/S clinic day to provide real-time teleultrasound mentorship. Clinician trainees scan the breast, document their independent findings and management plan in the study REDCap database, and then "call" the supervisor using Reacts. Reacts permits supervisor and trainee to see each other virtually; the supervisor can also view live U/S images and the trainee's probe and hand position to provide real-time feedback.
  Arms: Teleultrasound
Behavioral: Asynchronous virtual feedback — Clinicians at Arm 2 hospitals will save static images, with or without video at clinicians' discretion, onto the Philips Lumify tablets. These will be uploaded to a secure internet-based folder with case descriptions, and assigned U.S.- and Rwanda-based experts will be notified that images are available. Experts will review images within 24 hours and email feedback to trainees on imaging quality/ technique and management; trainees can also email questions.
  Arms: Asynchronous virtual feedback

SUMMARY:
Diagnosing breast cancer early is critical to reduce preventable breast cancer deaths in sub-Saharan Africa. This can be done in part through increasing patients' access to breast ultrasound, which is essential for evaluating breast masses. However, ultrasound is typically provided only by radiologists at urban referral hospitals. Training clinicians at rural district hospitals who are not radiologists could increase patients' access to breast ultrasound, but strategies to support and supervise these clinicians and ensure they are providing high-quality ultrasound services has not been studied.

This project will examine the effectiveness and cost of two strategies for training non-radiologist clinicians to perform breast ultrasound in Rwandan district hospitals.

DETAILED DESCRIPTION:
Breast cancer cases and deaths are rising rapidly in low- and middle-income countries (LMIC), including in sub-Saharan Africa, where most women with breast cancer are diagnosed with advanced-stage disease. Largely because of late-stage presentations, breast cancer survival in sub-Saharan Africa is poor. To address these global breast cancer inequities, the World Health Organization has emphasized the need for expanded access to breast cancer diagnostics in LMIC, and particularly calls for strategies that decentralize diagnostic testing to primary- and secondary-level health facilities while maintaining care quality. Diagnostic breast ultrasound (U/S) is an evidence-based intervention that is essential in evaluation of palpable breast abnormalities, including for determining which lesions require biopsy. However, diagnostic breast U/S is typically only provided by radiologists at LMIC referral facilities and is hard for low-income rural patients to access, impeding quality, equity, timeliness and efficiency of breast evaluation and contributing to diagnostic inefficiencies and delays. To address this issue, Rwanda's chief health implementation agency (Rwanda Biomedical Centre) has called for decentralized provision of breast U/S at district hospitals through task-shifting to non-radiologist clinicians. Supportive supervision is regarded as essential for successful task-shifting. However, scalable strategies for clinical supervision of non-radiologist clinicians to ensure sustained provision of high-quality decentralized breast ultrasound have not been investigated. The investigators' preliminary work training a small group of non-radiologist clinicians in Rwanda suggests that virtual support through electronically shared images and asynchronous feedback is feasible and potentially beneficial after intensive and prolonged in person training. However, supervision with real-time teleultrasound technology could be more effective in facilitating ultrasound provision and quality in a broader population of district hospital clinicians receiving shortened in-person training.

The objective of this research project is to compare 2 implementation strategies (teleultrasound supervision and asynchronous virtual feedback) to facilitate decentralized breast ultrasound at Rwandan district hospitals. The investigators will conduct a hybrid Type 2 implementation-effectiveness trial to accomplish this.

In Aim 1, the investigators will compare the strategies' impact on penetration of guideline-concordant diagnostic breast ultrasound at district hospitals (implementation effectiveness).

In Aim 2, the investigators will compare the strategies' impact on trainee-performed breast U/S image quality at district hospitals (clinical effectiveness).

In Aim 3, the investigators will estimate the implementation strategies' costs and cost-effectiveness in facilitating high-quality breast U/S, as well as examine downstream cost offsets associated with decentralized breast U/S.

These findings will directly inform breast cancer diagnosis pathways in Rwanda, shape the workforce and credentialing processes for breast U/S, and expand patients' access to this service. In addition, this project will contribute to global understanding of feasible, contextually appropriate and effective strategies to increase access to breast cancer diagnostic services (particularly imaging) in LMIC- a topic of major global interest in light of rapidly rising breast cancer incidence and mortality in LMIC.

ELIGIBILITY:
Enrollment in this cluster randomized clinical trial will occur at the health facility level.

Inclusion Criteria:

1. District hospital in Rwanda;
2. Already implementing the Women's Cancer Early Detection Program in their districts (i.e. clinicians in health centers and hospitals in the district have received the nationally-sponsored trainings in breast cancer early detection and cervical cancer screening);
3. Already using the WCEDP electronic medical record in health centers and the district hospital, or prepared to start using it.

Exclusion Criteria:

1. Already providing routine breast ultrasound in the district hospital.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1792 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Penetration of diagnostic breast ultrasound provision in district hospitals | 12 months
  Number of women receiving breast U/S / number of individuals evaluated at the district hospital with a breast mass
Trainee-provided breast ultrasound quality | 12 months
  Image quality score assessed by a blind third-party radiologist using a 15-item quality metric. Score is currently being validated and finalized.

SECONDARY OUTCOMES:
Fidelity to assigned clinical support implementation strategy | 12 months
  Out of total number of ultrasounds performed, % performed using the assigned clinical support strategy (teleultrasound or asynchronous feedback)
Adoption of breast U/S by clinicians | 12 months
  % of weeks in which ultrasound is provided
Maintenance of breast U/S provision | 13-24 months
  % of weeks that U/S is provided
Maintenance of breast U/S volume | 13-24 months
  Number of U/S scans per week
Feasibility of implementation strategies | Months 3,6,12
  4-item instrument measuring the feasibility of an intervention, included in clinician and site leadership surveys. Scores can range from 0-20, with higher scores indicating greater feasibility.
Appropriateness of implementation strategies | Months 3,6,12
  4-item measure of appropriateness of intervention, included in clinician and site leadership surveys. Score can range from 0-20. Higher scores indicate greater appropriateness.
Sustainment of implementation strategies | 24 months
  3-item Provider REport of Sustainment Scale (PRESS) included in clinician and leadership surveys. Each item is scored 0 = not at all, 1 = to a slight extent, 2 = to a moderate extent, 3 = to a great extent, and 4 = to a very great extent. Minimum score=0 (not sustained); maximum score=12 (sustained to a great degree).

CONTACTS AND LOCATIONS:
Overall Officials: Lydia E Pace, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners in Health (Inshuti Mu Buzima), Butaro, Rwanda

IPD SHARING:
Plan to Share IPD: No
Data sharing will only be implemented in accordance with Rwanda's data security regulations. No individual-level data will be shared.